CLINICAL TRIAL: NCT06688045
Title: A Study to Evaluate the Effects of Multiple Oral Doses of Itraconazole on the Single-dose Pharmacokinetics of Nemtabrutinib in Healthy Male Participants
Brief Title: A Study of the Effects of Itraconazole on the Plasma Levels of Nemtabrutinib (MK-1026-013)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 1026-013; MK-1026-013 (Other: MSD)
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: Healthy
MeSH Terms: interventions — ARQ531; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Period 1: Nemtabrutinib (Experimental): Participants receive a single oral dose of nemtabrutinib followed by a protocol specified wash-out period.
  Interventions: Drug: Nemtabrutinib
- Period 2: Nemtabrutinib + Itraconazole (Experimental): Participants receive oral doses of itraconazole once daily on Days 1 to 13 with a single oral dose of nemtabrutinib given with itraconazole on Day 4.
  Interventions: Drug: Nemtabrutinib; Drug: Itraconazole

INTERVENTIONS:
Drug: Nemtabrutinib — Oral administration
  Other Names: MK-1026; ARQ-531
Drug: Itraconazole — Oral administration
  Arms: Period 2: Nemtabrutinib + Itraconazole

SUMMARY:
The goal of this study is to learn what happens to levels of nemtabrutinib in a person's body over time. Researchers will compare what happens to nemtabrutinib in the body when it is given with or without another medicine called itraconazole.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health based on medical history, physical examination, vital sign (VS) measurements, electrocardiograms (ECGs) and laboratory safety tests performed before allocation.
* Has a body mass index (BMI) of18 to 32 kg/m^2 (inclusive)

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases.
* Has a history of cancer (malignancy).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Assigned male sex at birth.
Enrollment: 15 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-01-06 (Actual); Study Completion 2024-01-06 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Nemtabrutinib | At designated time points (up to approximately 10 days postdose)
  Blood samples will be collected to determine the AUC0-inf of nemtabrutinib in plasma.
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-last) of Nemtabrutinib | At designated time points (up to approximately 10 days postdose)
  Blood samples will be collected to determine the AUC0-last of nemtabrutinib in plasma.
Maximum Plasma Concentration (Cmax) of Nemtabrutinib | At designated time points (up to approximately 10 days postdose)
  Blood samples will be collected to determine the Cmax of nemtabrutinib in plasma.
Time of Maximum Plasma Concentration (Tmax) of Nemtabrutinib | At designated time points (up to approximately 10 days postdose)
  Blood samples will be collected to determine the Tmax of nemtabrutinib in plasma.
Apparent Terminal Half-life (t1/2) of Nemtabrutinib | At designated time points (up to approximately 10 days postdose)
  Blood samples will be collected to determine the t1/2 of nemtabrutinib in plasma.
Apparent Clearance (CL/F) of Nemtabrutinib | At designated time points (up to approximately 10 days postdose)
  Blood samples will be collected to determine the CL/F of nemtabrutinib in plasma.
Apparent Volume of Distribution (Vz/F) of Nemtabrutinib | At designated time points (up to approximately 10 days postdose)
  Blood samples will be collected to determine the Vz/F of nemtabrutinib in plasma.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 6 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue from Study Due to an AE | Up to approximately 6 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Labcorp Clinical Research Unit Inc. (Site 0001), Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/